CLINICAL TRIAL: NCT01055665
Title: Cognitive Behavioral Therapy, Self-Efficacy, and Depression in Persons With Chronic Pain
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virginia Nash, RN, Clinical Nurse Specialist, Mayo Clinic
Other Study IDs: 09-003969
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: cognitive behavior therapy — 6 cognitive behavior therapy groups

SUMMARY:
The investigators are exploring the role of Cognitive Behavioral Therapy (CBT), a treatment for depression, on self-efficacy (feeling empowered to accomplish a given task) and depression in persons with chronic pain and depression. Past research has shown that persons with chronic pain show improvement in self-efficacy and depression scores when they are using CBT. The Pain rehabilitation Center (PRC) at Mayo Clinic is adding CBT focused groups to better understand the role of CBT on self-efficacy and depression in persons with chronic pain and depression.

DETAILED DESCRIPTION:
Subjects will need to complete two questionnaires on admission and on discharge from the PRC program to measure self-efficacy and depression. The first is the Pain Self-Efficacy Scale (PSEQ) which is a measure of self-efficacy in persons with chronic pain. The second questionnaire is the Center for Epidemiologic Studies Depression Scale (CES-D) which is a measure of depressive symptoms in persons with chronic pain. Both scales will also be used for clinical information. Persons who score 27 or higher on the CES-D will be approached for potential consent to this evidence based project. Each patient in the PRC will participate in up to 6 CBT sessions but only persons who, upon admission, score 27 or greater on the CES-D will be studied for any changes in scores from admission to discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over with chronic pain and
* score of 27 or higher on CES-D scale

Exclusion Criteria:

* 17 or younger, no chronic pain,
* cognitively unable to participate in programming

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with chronic pain and depressive symptoms in a pain rehabilitation program.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change on a depression and self-efficacy scale | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Virginia R Nash, RN, MS, CNS, Principal Investigator — Mayo Clinic